CLINICAL TRIAL: NCT00091520
Title: Follow-up Serial Infusions of Natrecor(Nesiritide) in the Management of Patients With Heart Failure-FUSION II
Brief Title: A Study of the Safety and Efficacy of Follow-up Serial Infusions of Natrecor(Nesiritide) for the Management of Patients With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003355
Record Dates: First submitted 2004-09-09; First posted 2004-10-01 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2010-03

CONDITIONS: Heart Failure, Congestive
Keywords: Congestive heart failure; Nesiritide
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: Nesiritide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nesiritide administered as serial infusions to heart failure (HF) patients in the outpatient setting.

DETAILED DESCRIPTION:
Heart Failure (HF) is the inability of the heart to pump efficiently and the heart cannot perform the necessary circulation of blood through the body. This can result in symptoms like shortness of breath at rest or with minimal activity. Advanced heart failure is one of the leading causes of hospitalization and deaths in the United States. This is a prospective randomized, double-blind, placebo-controlled parallel group, multicenter study of the effectiveness of Nesiritide administered as serial infusions in the outpatient setting. Patients enrolled in this study will receive nesiritide or placebo for up to 12 weeks. Patients will then be followed for an additional 12 weeks. During the the first 17 weeks of the study patients will have multiple laboratory tests, have their vital signs (blood pressure and heart rate) assessed, and complete quality of life questionnaires. During the last few weeks of the study patients will be contacted to inquire how they are doing. The study hypothesis is that compared to placebo plus standard care, Nesiritide plus standard will reduce time to death or first occurrence of hospitalization due to heart or kidney problems. Safety will be assessed through the collection of adverse events, clinical laboratory tests and vital signs at various time points throughout the study. The patients assigned to the nesiritide group will receive a single 2.0mcg/kg bolus (one time injection) followed by serial IV infusions (4 to 6 hours) at a standard flow rate of 0.010 mcg/kg/min once or twice per week for 12 weeks. The patients assigned to the placebo group will receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Had at least two qualifying hospitalizations or hospitalization equivalents in the past year, with the most recent hospitalization or hospitalization equivalent within the past 60 days, but who has been out of the hospital at least 5 days (the day of discharge is day 0)
* Have documentation indicating that the patient was consistently New York Heart Association (NYHA) Class III or IV during the 60 days before randomization
* Have a Left Ventricular Ejection Fraction less than 40% (measured within 24 weeks before randomization)
* Are (1)NYHA Class IV or (2)NYHA Class III with highest calculated CrCl, 60mL/min within the previous 30 days
* Are receiving optimal treatment with long-term oral medications (e.g., diuretics, angiotensin converting enzyme (ACE) inhibitors, angiotensin II receptor blockers (ARBs), and beta blockers, unless these are documented to be contraindicated or not tolerated)
* Agree to come to the clinic up to 2 times per week (according to randomization) for 16 weeks of study drug infusions and to participate in all required follow-up assessments through week 24. In addition, agree to be contacted monthly after week 24 for follow-up, until the entire study has been completed

Exclusion Criteria:

* Have systolic blood pressure consistently <90mm Hg
* Are unable or unwilling to discontinue intermittent or continuous infusions of dopamine, dobutamine, milrinone, nitroglycerin, or open-label Natrecor beginning at the time of the screening visit
* Have required recent outpatient IV vasoactive (milrinone, dobutamine, dopamine, nitroglycerin, or open-label Natrecor) therapy as defined as >2 outpatient (excluding emergency room or inpatient) infusions in the last 30 days without a subsequent hospitalization
* Had, or during the course of the study are anticipated to have, any organ transplantation (heart, liver, lung, kidney, or bone marrow)
* Had a biventricular pacemaker placed within the 45 days before randomization or a single or dual chamber pacemaker or an automatic implantable cardiac defibrillator placed within the 15 days before randomization
* Have cardiogenic shock, volume depletion, or any other clinical condition at the time of randomization that would contraindicate the administration of Natrecor
* Are currently receiving chronic dialysis or have the expectation that dialysis will be required during the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2004-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to all-cause death or first occurrence of hospitalization for cardiovascular and/or renal causes from the day of randomization through week 12.

SECONDARY OUTCOMES:
Number of cardiovascular and/or renal hospital admissions adjusted for duration of observation period through the end of week 12. Days alive and out of the hospital from the day of randomization through the end of week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Derived] Yancy CW, Krum H, Massie BM, Silver MA, Stevenson LW, Cheng M, Kim SS, Evans R; FUSION II Investigators. Safety and efficacy of outpatient nesiritide in patients with advanced heart failure: results of the Second Follow-Up Serial Infusions of Nesiritide (FUSION II) trial. Circ Heart Fail. 2008 May;1(1):9-16. doi: 10.1161/CIRCHEARTFAILURE.108.767483. PMID 19808265
- See also: Follow-up Serial Infusions of Natrecor(Nesiritide) in the Management of Patients With Heart Failure-FUSION II — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=955&filename=CR003355_CSR.pdf